CLINICAL TRIAL: NCT00366691
Title: Comparison of Acular LS With Lotemax to Prevent Anterior Segment Inflammation After Phacoemulsification and Intraocular Lens Implantation
Brief Title: Comparison of Acular LS With Lotemax to Prevent Inflammation After Cataract Surgery and Intraocular Lens Implantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRC-06-002
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2006-06

CONDITIONS: Cataract Extraction
Keywords: cataract
MeSH Terms: conditions — Cataract | interventions — Ketorolac; Loteprednol Etabonate

INTERVENTIONS:
Drug: Acular LS
Drug: Lotemax

SUMMARY:
The purpose of this study is to compare the effectiveness of Acular LS® and Lotemax® in the prevention of inflammation in the eye after cataract surgery. Acular LS is made by Allergan, Inc. It is a nonsteroidal anti-inflammatory drug (NSAID) and is approved by the Food and Drug Administration (FDA) for use following cataract surgery. Lotemax is made by Bausch & Lomb. It is a steroid and is also approved by the FDA for use following cataract surgery.

DETAILED DESCRIPTION:
Ketorolac tromethamine is a nonsteroidal anti-inflammatory drug (NSAIDs) which, when administered systemically, has demonstrated analgesic, anti-inflammatory, and anti-pyretic activity. The mechanism of its action is thought to be due to its ability to inhibit prostaglandin biosynthesis (cyclo-oxigenase inhibitors). However, they leave the lipoxygenase pathway free to generate leukotrienes. This pharmacodynamic activity has been speculated as a reason why NSAIDs produce less ocular side effects than corticosteroids. It has been widely used in ophthalmology. In 1987, Flach1 published its effectiveness in the treatment of aphakic and pseudophakic macular edema. Its efficacy after cataract surgery has been shown2 and it has been compared to topical steroids after extra-capsular cataract extraction3,4,5 and phacoemulsification6,7. It has been used as analgesic after radial keratotomy(RK)8,9, photorefractive keratectomy (PRK)10 and laser in situ keratomileusis (LASIK)11

The purpose of this study is to compare the effectiveness of the NSAID ketorolac tromethamine ophthalmic solution 0.4% with the steroid loteprednol etabonate ophthalmic suspension 0.5% for preventing anterior segment inflammation after routine cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a visually significant age-related cataract, in the planned operated eye.
* 18 years of age or older.
* The vision in the fellow, unoperated eye should have a potential visual acuity of 20/40 or better as determined by the principal investigator.
* Patient must desire cataract extraction.
* Willing and able to comply with scheduled visits and other study procedures.

Exclusion Criteria:

* Advanced glaucomatous damage.
* Any abnormality preventing reliable applanation tonometry in operated eye.
* Contact lens use during the active treatment portion of the trial in the operated eye.
* Any concurrent infectious/non infectious conjunctivitis, keratitis or uveitis in either eye.
* Any history of allergic hypersensitivity or poor tolerance to any component of the preparations used in this trial.
* Pregnant or nursing mothers and females of childbearing potential not practicing a reliable and medically acceptable method of birth control.
* Any clinically significant, serious or severe medical or psychiatric condition.
* Participation in (or current participation) any investigational drug or device trial within the previous 30 days prior to the start date of this trial.
* Intraocular conventional surgery within the past three months or intraocular laser surgery within one month in the operated eye.
* Required use of other topical medications during the active portion of the trial except prophylactic antibiotic, topical lid care, tear replacement solutions or glaucoma medications.
* Other ocular surgery at the time of the cataract extraction.
* Use of topical or oral antiprostaglandins or corticosteroids as well as aspirin products (> 81 mg) during the active treatment portion of the trial. If patient wants to participate in the trial and can stop the medication, he/she can be enrolled after 7-day wash out period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2006-02; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry D Solomon, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Storm Eye Institute, Medical University of South Carolina, Charleston, South Carolina, United States